CLINICAL TRIAL: NCT04260529
Title: A First-in-human, Open-label Dose Escalation Followed by Dose Expansion Phase I/IIa Trial to Evaluate the Safety, Preliminary Efficacy and Pharmacokinetics of Intratumoral CyPep-1 Monotherapy and in Combination With Pembrolizumab in Patients With Advanced Solid Cancers.
Brief Title: CyPep-1 Injections in Cancer Inducing Lymphocyte Infiltrate Accumulations
Acronym: CICILIA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytovation AS (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CyPep-1; 2019-003317-33 (EudraCT Number); KEYNOTE-D02 (Other: Merck Sharp & Dohme LLC); MK-3475-D02 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor Malignancy
Keywords: Cancer; Tumour; Oncology; Immunotherapy; Oncolytic; Cluster of Differentiation 8 (CD8)); Intratumoral; Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Phase I Cohort 1 (Experimental): Dose escalation at 0.5 mg (milligrams)/mL, n=3
  Interventions: Drug: CyPep-1
- Phase I Cohort 2 (Experimental): Dose escalation at 2 mg/mL, n=5
  Interventions: Drug: CyPep-1
- Phase I Cohort 3 (Experimental): Dose escalation at 5 mg/mL, n=6
  Interventions: Drug: CyPep-1
- Phase IIa: Arm A (Experimental): CyPep-1 5.0mg/mL Monotherapy
  Interventions: Drug: CyPep-1
- Phase IIa Arm B (Experimental): The safety and tolerability of CyPep-1 in combination with pembrolizumab was evaluated in a cohort of 15 patients in total, using a staggered approach. Initially, 3 patients received CyPep-1 at Recommended Phase 2 Dose (RP2D) in combination with pembrolizumab once every 6 weeks (Q6W)
  Interventions: Drug: CyPep-1; Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®]
- Phase IIa Arm C Cohort 4 (Experimental): The safety and tolerability of at least 2 dose levels of CyPep-1, the RP2D and the dose immediately below that, were evaluated when CyPep-1 was administered IT using ultrasound guidance to one metastatic lesion in the liver (Cohort 4: 2 mg/mL, n=6)
  Interventions: Drug: CyPep-1
- Phase IIa Arm C Cohort 5 (Experimental): The safety and tolerability of at least 2 dose levels of CyPep-1, the RP2D and the dose immediately below that, were evaluated when CyPep-1 was administered intratumoral (IT) using ultrasound guidance to one metastatic lesion in the liver. The RP2D (Cohort 5: 5 mg/mL, n=6).
  Interventions: Drug: CyPep-1
- Phase IIa Arm D (Experimental): The safety and tolerability of CyPep-1 at RP2D was planned to be further evaluated with focus on assessing efficacy signals of CyPep-1 monotherapy in 30 patients with cutaneous melanoma.
  Interventions: Drug: CyPep-1

INTERVENTIONS:
Drug: CyPep-1 — Intratumoral injection
Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®] — IV infusion
  Other Names: KEYTRUDA®
  Arms: Phase IIa Arm B

SUMMARY:
This Phase I/IIa trial is designed to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of CyPep-1 when administered directly into malignant tumors in monotherapy and in combination with anti programmed cell death protein 1(anti-PD-1) antibody pembrolizumab. Additionally, the trial will monitor anti-tumor effects on both injected lesions and distant non-injected deposits.

DETAILED DESCRIPTION:
Treatment with immune modulating agents may result in long lasting anti-tumor responses in patients with cancer. However, only a subset of patients obtains durable remission. Treatment strategies that aim at recruiting tumor antagonizing cellular components of the immune system holds great promise. CyPep-1 is a chemically synthesized peptide with oncolytic properties. It selectively targets cancer cells based on their altered molecular composition, and removes the surrounding cell membrane. This releases tumor neoantigens to the microenvironment and potentially induces an anti-tumour immune response.

Preclinical studies showing that CyPep-1 can synergize with anti-PD-1 antibody treatment in terms of decreased tumor volumes and prolonged survival highlight the possible clinical utility of CyPep-1 in the combination setting with Immune checkpoint inhibitors (ICIs).

This is a phase I/IIa, open label trial, with a dose escalation phase to evaluate the safety and tolerability of CyPep-1 as monotherapy and in combination with pembrolizumab, to identify the recommended phase 2 dose, followed by a dose expansion phase in subjects with advanced solid tumors. The trial consists of two phases and multiple arms.

Secondary objectives are preliminary anti-tumor efficacy and to assess the pharmacokinetics (PK) of CyPep-1 as monotherapy and in combination with pembrolizumab. As part of the exploratory analysis, it is planned to determine local and systemic immunological effects after CyPep-1 administration, alone and in combination with pembrolizumab.

ELIGIBILITY:
Inclusion criteria:

For Phase I and Phase IIa Arms A and C:

1. Histologically or cytologically confirmed locally advanced (unresectable) or metastatic tumors (solid tumor or lymphoma) with an accessible tumor lesion for intratumoral injection of CyPep-1 malignancy (including lymphomas) that is either:

   1. Refractory to standard-of-care treatment
   2. Have a disease for which there is no standard therapy considered appropriate. Metastatic deposits (including cutaneous/subcutaneous lesions and metastatic deposits in lymph nodes) of tumors for which IT injections may be performed are eligible. Pure cutaneous infiltrations (e.g., breast cancer cutaneous carcinomatosis) are ineligible.
2. 1 to 3 non-ulcerated transcutaneously accessible lesion(s) for injection and measurable as defined by Immune Response Evaluation Criteria in Solid Tumors (iRECIST). All other tumor lesion(s) may be selected for efficacy follow-up but will not be subjected to treatment with CyPep-1.
3. Presence of tumor lesion(s) (that have not been previously irradiated) suitable for biopsy at screening and at Week 6.

   For Arm C:
4. Confirmation of the presence of at least 1 liver metastasis by imaging.
5. Subjects must have measurable disease which is equal to one or more metastatic liver lesions that can be accurately and serially measured that are greater than 1 cm dimension and for which the longest diameter is greater or equal to 1 cm as measured by computed tomography (CT) scan or magnetic resonance imaging (MRI). The metastatic liver lesion must not be in an area that received prior localized therapies.
6. Metastatic liver lesion for injection with >50% radiological visible necrosis must be avoided and the lesion must be located where any tumor swelling will not lead to gall bladder tract obstruction or lead to bleeding risk.

   For Arm D:
7. Histologically or cytologically confirmed diagnosis of advanced (unresectable Stage III) or metastatic (Stage IV: M1a) melanoma considered incurable by Standard of Care. For metastatic melanoma, only distal cutaneous, subcutaneous, or lymph node metastases are allowed.
8. Previously exposed to ICI(s) and be categorized following the Society for Immunotherapy of Cancer (SITC) Immunotherapy Resistance Taskforce meeting one of the following:

   a. Have primary resistance: PD-(L)-1 inhibitor exposure ≥6 weeks and have the best response as one of the following: i. Progressive disease/ Disease progression (PD), ii. Stable Disease (SD) for <6 months. b. Have secondary resistance: PD-(L)-1 inhibitor exposure ≥6 weeks and best response Complete response (CR), Partial Response (PR), or SD >6 months.

   c. Have adjuvant therapy resistance: recurrence subcategorized into primary resistance/early relapse occurred <12 weeks after the last dose, and late relapse occurred ≥12 weeks after the last dose. If B-Raf gene (BRAF) mutated, patients must have progressed to treatment with BRAF inhibitors.

   d. Have neoadjuvant therapy resistance including subjects with or without major pathologic response and subsequent PD that fulfills criteria for primary or secondary resistance e. Discontinued from ICI(s) therapy due to immune-related adverse events grade 3 or 4 other than endocrine insufficiencies treatable with hormonal replacement therapy, and meet one of the following: i. Remain on SD at discontinuation of PD-(L)1 inhibitor in combination with ipilimumab or show regrowth after <12 weeks of the last dose ii. Have not achieved a CR with single-agent PD-(L)1 inhibitor or combination of PD-(L)1 with Lymphocyte activation gene-3 (LAG-3) inhibitor
9. At least 1 non-ulcerated lesion, not exceeding 5 cm in (the longest) diameter, for intratumoral injection(s) and measurable as defined by iRECIST.
10. Resolution of toxicity due to prior therapy returned to baseline or < Grade 2, except for alopecia or other irreversible immune-mediated AEs, as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. and SITC ICI-related Adverse events (AEs).
11. Prior treatment(s) delivered by IT injection to the to-be injected lesion(s), including investigational agents, is allowed.

    For Phase I and Phase IIa Arms A, C, and D in addition:
12. Age ≥ 18 years.
13. Estimated life expectancy of at least 3 months.
14. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
15. Resolution of toxicity due to prior therapy to Grade < 2 (except for alopecia and transaminases in case of liver metastases) as defined by CTCAE v5.0.
16. Ability to give written informed consent and to comply with the protocol.
17. All subjects of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must have a negative highly sensitive pregnancy test at screening (urine/serum) and agree to use highly effective method for contraception according to the European Union (EU) Clinical Trial Facilitation Group guidance from time of signing the informed consent form (ICF) until at least 120 days after the last administration of CyPep-1. The partners of subjects with childbearing potential must also apply contraceptive methods and are recommended not to donate sperm.
18. Adequate bone marrow, liver, and renal function:

    1. Platelet count ≥ 100 x 109/L
    2. Hemoglobin ≥ 6.0 mmol/L or 9.67 g/dL
    3. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
    4. Total bilirubin ≤ 1.5 x Upper limit of normal (ULN), except for subjects with familial bilirubinemia (Gilbert's disease)
    5. Serum Aspartate transaminase (ASAT) and Alanine transaminase (ALAT) ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastases)
    6. Creatinine clearance ≥ 30 mL/min (by CKD-EPI formula).

    For Phase IIa Arm B:

    Participants are eligible to be included in Arm B of the trial only if all of the following criteria apply:
19. The participant provides written informed consent for the trial.
20. Be ≥ 18 years of age on day of signing informed consent.
21. Participant with histologically or cytologically confirmed diagnosis of advanced (unresectable Stage III) or metastatic (Stage IV) solid tumor malignancy (including lymphomas) that is refractory to standard-of-care treatment or for which there is no standard therapy considered appropriate. Metastatic deposits (including cutaneous/subcutaneous lesions and metastatic deposits in lymph nodes) of tumors for which IT injections may be performed are eligible. Pure cutaneous infiltrations (e.g., breast cancer cutaneous carcinomatosis) are ineligible.
22. Subjects must have progressed on treatment with an anti-Programmed cell death protein 1 (PD1)/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. Treatment progression is defined by meeting all of the following criteria:

    1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
    2. Has demonstrated clinical or radiological disease progression (PD) after PD-1/L1
23. A male participant must agree to use contraception and refrain from sperm donation during the treatment period and for at least 120 days after the last dose of trial medication.
24. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP)
    2. A WOCBP (defined as < 2 years after last menstruation or not surgically sterile) must have a negative highly sensitive pregnancy test at screening (urine/serum) and must follow contraceptive guidance (highly effective method for contraception according to the EU Clinical Trial Facilitation Group guidance) from time of signing the ICF until at least 120 days after the last administration of trial medication. The partners of subjects with childbearing potential must also apply contraceptive methods and are recommended not to donate sperm.
25. 1 to 3 non-ulcerated transcutaneously accessible lesion(s) for injection and measurable as defined by iRECIST. All other tumor lesion(s) may be selected for efficacy follow-up but will not be subjected to treatment with CyPep-1.
26. Presence of tumor lesion(s) (that have not been previously irradiated) suitable for biopsy at screening and at Week 6.
27. Have an ECOG performance status of 0 to 1.
28. Have adequate organ function as defined in the following table. Specimens must be collected within 10 days (or less) prior to the start of trial treatment.
29. Only for subjects with lymphoma: have measurable disease defined as at least one lesion that can be accurately measured in at least two dimensions with spiral CT scan. Minimum measurement must be > 15 mm in the longest diameter by > 10 mm in the short axis.
30. Estimated life expectancy of at least 3 months.
31. Human immunodeficiency virus (HIV) infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease.

Exclusion criteria:

For Phase I and Phase IIa Arms A, C, and D: subjects who meet any of the following criteria at screening will be excluded from trial entry:

1. There is no limit to the number of prior treatment regimens, but prior treatment(s) should not include compounds delivered by IT injection to the to-be injected lesion(s), including investigational agents. Subjects with prior IT therapies are allowed in Arm D.
2. Participation in another clinical trial within 4 weeks prior to first dose of CyPep-1.
3. Anti-cancer therapy within 4 weeks prior to the first dose of CyPep-1 (within 2 weeks for palliative radiotherapy, within 1 week for endocrine therapy).
4. Major surgical procedure within 14 days prior to the first dose of CyPep-1.
5. Live vaccine within 30 days prior to first dose of CyPep-1.
6. Expected to require any other form of systemic or localized antineoplastic therapy while in this trial. Localized palliative radiotherapy for pain relief is allowed on tumor lesions that are not selected for evaluation of treatment response.
7. Clinical evidence of an active second malignancy that is progressing or requires active treatment, except for curatively treated early stage (carcinoma in situ or stage 1) carcinomas or non-melanoma skin cancer.
8. Active autoimmune disease requiring immunosuppressive therapy.
9. Any condition requiring continuous systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive agents within 2 weeks prior to first dose of CyPep-1. Inhaled, intranasal or topical (only on areas outside the injected lesion[s]) and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active auto-immune disease.
10. Abnormal or clinically significant coagulation parameters:

    1. Prothrombin Time - International Normalized Ratio (PT-INR) ≥ 1.5 ULN
    2. Activated Partial Thromboplastin Time (APTT) ≥ 1.5 ULN Subjects being treated with anticoagulants are excluded if the coagulation parameters are outside the therapeutic intervals as described in the Summary of Product Characteristics (SmPC) for the administered treatment.
11. Subjects on anticoagulants with temporarily stop and start, supported by low molecular weight heparin (or other anticoagulation therapy at the discretion of the investigator and/or per local standard of care) during treatment period.
12. Known hypersensitivity to any component of CyPep-1.
13. Prior allogeneic tissue/solid organ transplant, stem cell or bone marrow transplant.
14. Known active human immunodeficiency virus (HIV). Subject is eligible when normal levels of Cluster of Differentiation 4 (CD4) are present.
15. Central nervous system (CNS) metastasis that is symptomatic or progressing or that requires current therapy (e.g., evidence of new or enlarging CNS metastasis, carcinomatous meningitis or new neurological symptoms attributable to CNS metastasis).
16. QTcF (QT corrected for heart rate by Fridericia's cube root formula)> 480 ms, history of long or short QT syndrome, Brugada syndrome, or known history of QTc (Corrected QT Interval) prolongation, or Torsade de Pointes.
17. Women who are pregnant or breastfeeding.
18. Any serious and/or unstable pre-existing medical, psychiatric or other condition which in the investigator's opinion could interfere with subject safety, obtaining written informed consent, or compliance with the trial protocol.

    Additional exclusion criteria for Phase IIa Arm C:
19. Subject is a candidate for hepatic surgery or local regional therapy of liver metastases with curative intent.
20. More than one third of the liver is estimated to be involved with metastases.
21. There is invasion by cancer into the main blood vessels such as the portal vein, hepatic vein or the vena cava.
22. Subject is currently receiving or has received liver metastatic-directed therapy (eg: radiation, ablation, embolization) less than 4 weeks prior to enrolment or hepatic surgery.

    Exclusion criteria specific for Phase IIa Arm B:

    Participants are excluded from the trial if ANY of the following criteria apply at screening:
23. A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to trial treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
24. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., Cytotoxic T-lymphocyte-associated protein (CTLA) 4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE).
25. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks (within 1 week for endocrine therapy) prior to first dose of CyPep-1.
26. Has received prior (palliative) radiotherapy within 2 weeks of start of trial treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
27. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of CyPep-1. Note: Administration of killed vaccines are allowed.
28. Has received prior compounds delivered by IT injection to the to-be injected lesion(s), including investigational agents.
29. Expected to require any other form of systemic or localized antineoplastic therapy while in this trial. Localized palliative radiotherapy for pain relief is allowed on tumor lesions that are not selected for evaluation of treatment response.
30. Ongoing pembrolizumab-related toxicity event(s) as per Treatment Limiting Toxicity (TLT) definition.
31. Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.
32. Has had an allogeneic tissue/solid organ transplant.
33. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of CyPep-1.
34. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years, except for curatively treated early stage (carcinoma in situ or stage 1) carcinomas or non-melanoma skin cancer.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
35. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
36. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients or to another mAb, as well as any known hypersensitivity to any component of CyPep-1.
37. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
38. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
39. Has an active infection requiring systemic therapy.
40. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
41. Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as Hepatitis C virus (HCV) RNA [qualitative] is detected) infection.
42. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
43. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
44. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of trial treatment (applicable only for subjects with non-small cell lung cancer [NSCLC], mesothelioma and small cell lung cancer [SCLC]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- France (2):
  - Institue Curie, Paris
  - Institute Gustave Roussy, Villejuif
- Netherlands (4):
  - NKI/AvL, Amsterdam
  - LUMC, Leiden
  - EMC, Rotterdam
  - UMCU, Utrecht
- Spain (2):
  - Vall d'Hebron (VHIO), Barcelona
  - START, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of study completion

REFERENCES:
- [Background] Gibney GT, Weiner LM, Atkins MB. Predictive biomarkers for checkpoint inhibitor-based immunotherapy. Lancet Oncol. 2016 Dec;17(12):e542-e551. doi: 10.1016/S1470-2045(16)30406-5. PMID 27924752
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Samstein RM, Lee CH, Shoushtari AN, Hellmann MD, Shen R, Janjigian YY, Barron DA, Zehir A, Jordan EJ, Omuro A, Kaley TJ, Kendall SM, Motzer RJ, Hakimi AA, Voss MH, Russo P, Rosenberg J, Iyer G, Bochner BH, Bajorin DF, Al-Ahmadie HA, Chaft JE, Rudin CM, Riely GJ, Baxi S, Ho AL, Wong RJ, Pfister DG, Wolchok JD, Barker CA, Gutin PH, Brennan CW, Tabar V, Mellinghoff IK, DeAngelis LM, Ariyan CE, Lee N, Tap WD, Gounder MM, D'Angelo SP, Saltz L, Stadler ZK, Scher HI, Baselga J, Razavi P, Klebanoff CA, Yaeger R, Segal NH, Ku GY, DeMatteo RP, Ladanyi M, Rizvi NA, Berger MF, Riaz N, Solit DB, Chan TA, Morris LGT. Tumor mutational load predicts survival after immunotherapy across multiple cancer types. Nat Genet. 2019 Feb;51(2):202-206. doi: 10.1038/s41588-018-0312-8. Epub 2019 Jan 14. PMID 30643254
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Szczepanski C, Tenstad O, Baumann A, Martinez A, Myklebust R, Bjerkvig R, Prestegarden L. Identification of a novel lytic peptide for the treatment of solid tumours. Genes Cancer. 2014 May;5(5-6):186-200. doi: 10.18632/genesandcancer.18. PMID 25061502
- [Background] Vesely MD, Schreiber RD. Cancer immunoediting: antigens, mechanisms, and implications to cancer immunotherapy. Ann N Y Acad Sci. 2013 May;1284(1):1-5. doi: 10.1111/nyas.12105. PMID 23651186
- [Background] Zappasodi R, Merghoub T, Wolchok JD. Emerging Concepts for Immune Checkpoint Blockade-Based Combination Therapies. Cancer Cell. 2018 Apr 9;33(4):581-598. doi: 10.1016/j.ccell.2018.03.005. PMID 29634946
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Cohort 1: 0,5 mg/mL CyPep-1 (max 4mL) every 2 weeks (Q2W)
- Phase I Cohort 2: 2 mg/mL CyPep-1 (max 4mL) Q2W
- Phase I Cohort 3: 5 mg/mL CyPep-1 (max 4mL) Q2W
- Phase IIa Arm A: 5 mg/mL CyPep-1 (max 4mL) Q2W, monotherapy
- Phase IIa Arm B: 5 mg/mL CyPep-1 (max 4mL) Q2W in combination with pembrolizumab 600mg every 6 weeks (Q6W)
- Phase IIa Arm C Cohort 4: 2 mg/mL CyPep-1 (max 4mL) Q2W for liver metastases
- Phase IIa Arm C Cohort 5: 5 mg/mL CyPep-1 (max 4mL) Q2W for liver metastases
- Phase IIa Arm D: 5 mg/mL CyPep-1 (max 4mL) every week for 16 weeks for melanoma
Period: Overall Study
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
Started | 3 | 5 | 6 | 18 | 15 | 6 | 6 | 1
Completed | 3 | 5 (One participant withdrew consent.) | 6 | 18 | 15 | 6 | 6 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase IIa Arm D: 5 mg/mL CyPep-1 weekly for 16 weeks for melanoma
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D | Total
Number analyzed (Participants) | 3 | 5 | 6 | 18 | 15 | 6 | 6 | 1 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.2) | 64.6 (10.8) | 57.7 (5.9) | 57.9 (11.9) | 63.3 (8.4) | 64.0 (8.8) | 59.5 (13.7) | 55 (0) | 60.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 11 | 7 | 4 | 3 | 0 | 30
  Male | 2 | 3 | 4 | 7 | 8 | 2 | 3 | 1 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG [Count of Participants; unit: Participants] — Measure Description: Participants were eligible for the study with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry on all pre-disease performance without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work).
  Participants
    Grade 0 | 0 | 1 | 2 | 6 | 4 | 3 | 2 | 0 | 18
    Grade 1 | 3 | 4 | 4 | 12 | 11 | 3 | 4 | 1 | 42

OUTCOME MEASURES:

1. Primary Outcome: Type and Number of Adverse Events (AEs)
Description: According to National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) criteria v5.0, and additional safety parameters.
Time Frame: From Informed Consent Form (ICF) signing until Follow Up (FU) or until End of Treatment (EoT) visit. After FU visit, only ongoing AEs or Serious Adverse Events (SAEs) related to CyPep-1 were collected. Duration: up to a maximum of 28 months.
Measure: Number; unit: number of events
Groups:
- Phase I Cohort 1: 0.5 mg/mL CyPep-1 (max 4 mL) every 2 weeks (Q2W)
- Phase I Cohort 2: 2 mg/mL CyPep-1 (max 4 mL) Q2W
- Phase I Cohort 3: 5 mg/mL CyPep-1 (max 4 mL) Q2W
- Phase IIa Arm A: 5 mg/mL CyPep-1 (max 4 mL) Q2W, monotherapy
- Phase IIa Arm B: 5 mg/mL CyPep-1 (max 4 mL) Q2W in combination with pembrolizumab 600mg every 6 weeks (Q6W)
- Phase IIa Arm C Cohort 4: 2 mg/mL CyPep-1 (max 4 mL) Q2W for liver metastases
- Phase IIa Arm C Cohort 5: 5 mg/mL CyPep-1 (max 4 mL) Q2W for liver metastases
- Phase IIa Arm D: 5 mg/mL CyPep-1 (max 4 mL) weekly for 16 weeks for melanoma
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
Number analyzed (Participants) | 3 | 5 | 6 | 18 | 15 | 6 | 6 | 1
number of events
  Treatment Emergent Adverse Event (TEAE) | 24 | 37 | 62 | 143 | 262 | 91 | 91 | 4
  TESAE | 1 | 0 | 0 | 3 | 7 | 1 | 3 | 0
  CTCAE Grade >= 3 | 9 | 4 | 5 | 8 | 12 | 4 | 12 | 0
  TEAE leading to Study Treatment discontinuation | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  TEAE leading to CyPep-1 interruption | 1 | 1 | 1 | 10 | 8 | 1 | 2 | 0
  TEAE leading to pembrolizumab interruption | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Dose limiting toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Treatment limiting toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: 28 days after the date of the initial response, defined by complete response (disappearance of all target lesions) and partial responses (>=30% decrease in the sum of the longest diameter of target lesions), according to Immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Time Frame: up to approximately 28 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with BOR iCR/iPR
Groups:
- Phase I Cohort 1: 0,5 mg/mL CyPep-1 (max 4 mL) every 2 weeks (Q2W)
- Phase IIa Arm B: 0,5 mg/mL CyPep-1 (max 4 mL) Q2W in combination with pembrolizumab 600mg every 6 weeks (Q6W)
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
Number analyzed (Participants) | 3 | 5 | 6 | 18 | 15 | 6 | 6 | 1
percentage of subjects with BOR iCR/iPR | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 21.8] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 97.5]

3. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as increase in the sum of diameters of target lesion(s) identified at baseline to >20% and >5 mm from nadir; unequivocal progression of non-target lesion(s) identified at baseline; and development of new lesion(s).
Time Frame: time from treatment start until disease relapse or disease progression (based on all lesions, using iRECIST) or death due to any cause, whichever occurred earliest (up to a maximum of 28 months)
Measure: Median (Full Range); unit: Months
Groups:
- Phase IIa Arm B: 5 mg/mL CyPep-1 (max 4 mL) Q2W in combination with pembrolizumab 600 mg every 6 weeks (Q6W)
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
Number analyzed (Participants) | 3 | 5 | 6 | 18 | 15 | 6 | 6 | 1
Months | 1.6 [1.2 to 1.9] | 1.4 [0.0 to 9.3] | 2.8 [1.6 to 12.3] | 1.8 [0.0 to 5.4] | 1.9 [0.6 to 12.9] | 2.1 [1.4 to 5.7] | 1.9 [1.8 to 16.6] | 0.0 [0.0 to 0.0]

4. Other Pre Specified Outcome: Overall Survival (OS)
Time Frame: from start of study treatment to the date of death with a maximum of 28 months
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
Number analyzed (Participants) | 3 | 5 | 6 | 18 | 12 | 6 | 6 | 1
Months | 5.2 [2.1 to 21.9] | 5.5 [0.6 to 16.6] | 13.2 [5.3 to 19.8] | 7.7 [1.0 to 26.2] | 5.8 [1.5 to 26.7] | 8.3 [3.3 to 26.3] | 4.2 [2.5 to 17.6] | 0.7 [0.0 to 0.7]

ADVERSE EVENTS:
Time Frame: Subjects will be monitored for AEs and Events of Clinical Interest (ECIs) from the time of ICF signature until the FU visit (or until EoT, if it occurs more than 30 days after the last CyPep-1 administration). After the FU or EoT visit, only ongoing AEs or SAEs related to CyPep-1 administration will be collected for up to a maximum of 28 months.
Groups:
- Phase I Cohort 1: 0.5 mg/mL CyPep-1 (max 4 mL) Q2W
- Phase IIa Arm B: 5 mg/mL CyPep-1 (max 4 mL) Q2W in combination with pembrolizumab 600 mg Q6W
Arm/Group | Phase I Cohort 1 | Phase I Cohort 2 | Phase I Cohort 3 | Phase IIa Arm A | Phase IIa Arm B | Phase IIa Arm C Cohort 4 | Phase IIa Arm C Cohort 5 | Phase IIa Arm D
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/5 | 6/6 | 13/18 | 14/15 | 5/6 | 5/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/5 | 0/6 | 3/18 | 2/15 | 1/6 | 2/6 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 6/6 | 18/18 | 15/15 | 6/6 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 (N=3) | Phase I Cohort 2 (N=5) | Phase I Cohort 3 (N=6) | Phase IIa Arm A (N=18) | Phase IIa Arm B (N=15) | Phase IIa Arm C Cohort 4 (N=6) | Phase IIa Arm C Cohort 5 (N=6) | Phase IIa Arm D (N=1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 (N=3) | Phase I Cohort 2 (N=5) | Phase I Cohort 3 (N=6) | Phase IIa Arm A (N=18) | Phase IIa Arm B (N=15) | Phase IIa Arm C Cohort 4 (N=6) | Phase IIa Arm C Cohort 5 (N=6) | Phase IIa Arm D (N=1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 3 (8) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 4 (6) | 6 (23) | 15 (58) | 12 (71) | 5 (15) | 5 (26) | 1 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 3 (5) | 9 (13) | 8 (15) | 2 (5) | 5 (6) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4) | 2 (14) | 5 (8) | 7 (11) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (3) | 5 (5) | 5 (6) | 2 (2) | 3 (3) | 0 (0)
Decrease appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (7) | 2 (4) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (5) | 2 (2) | 2 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 5 (9) | 2 (8) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Malaiase (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (4) | 1 (1) | 5 (7) | 3 (6) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment of Arm D was stopped after the inclusion of 1 subject, as recruitment of arm D was not feasible in the current environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04260529/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04260529/SAP_001.pdf